CLINICAL TRIAL: NCT02068274
Title: Continuous Monitoring of Patients Treated With Opioids for Chronic Pain and Its Impact on Patient Safety. A Feasibility Trial.
Brief Title: CO2 Monitoring Study
Status: Completed | Type: Observational
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Chief of University Internal medicine Clinic, Cantonal Hosptal, Baselland
Other Study IDs: 194/12
Record Dates: First submitted 2014-02-14; First posted 2014-02-21 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Chronic Pain; Hypercapnia; Quality of Life
MeSH Terms: conditions — Chronic Pain; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic pain: CO2 monitoring in chronic pain patients who treated with opioids.

SUMMARY:
Opioids are an effective instrument for patients with acute and chronic pain. Their route of administration ranges from transdermal to subcutaneous application through to Intravenous Patient-Controlled Analgesia (IV-PCA).

The use of IV-PCA-pumps has considerable advantages including decreased delay in the administration of opioids from the time requested, individual dose intervals, self -control of their therapy, rapidity and ease of dose titration . These potential benefits, however are balanced by the need for careful assessment of adverse effects, including decreased quality of life because of the patient's sedation, constipation and possible episodes of bradypnoea and desaturation, eventually leading to respiratory depression (RD) requiring treatment. Often described safety features that help prevent overdosing are PCA bolus dose, delay, and lockout interval.

Even though the risk of serious, potentially life threatening complications by using IV-PCA without a background infusion was described to be very low (0.24%) compared to other methods of opioid delivery , adverse effects like worrying degrees of hypoxemia and bradypnoea do occur and often remain undetected due to the lack of continuous monitoring. One of the possible causes of patient harm are medication errors associated with PCA administration, a common form of PCA errors, which is a significant source of preventable patient morbidity and hospital resource utilization.

The individual patient response to a particular dose of opioids depends on diagnosed or unrecognized comorbidities. Clinical experience has shown that it is not possible to prospectively identify all patients who may be at increased risk.

Conventional opioid monitoring protocol may fail to detect frequent episodes of bradypnoea and desaturation measured by the respiratory rate (RR) and Saturation of Peripheral Oxygen (SpO2) because even at a low respiratory rate SpO2 is usually maintained, so that pulse oxymetry might fail to detect respiratory deterioration, particularly if a patient is receiving supplemental oxygen.

Therefore, continuous monitoring could be considered more sensitive, especially if it contains the measurement of Partial Pressure of Carbon dioxide (PCO2), which is a good parameter for monitoring ventilatory function.

The 'gold standard' method to measure the arterial partial pressure of carbon dioxide (PaCO2) is still the arterial blood gas analysis. But arterial sampling including catheterization or intermittent arterial puncture is invasive and expensive and associated with pain and discomfort for the patient. Therefore cutaneous carbon dioxide tension (PcCO2) measurement was suggested to be used as a non-invasive surrogate measure of PaCO2.

SpO2, and tcPCO2, are important clinical parameters that should be used in conjunction with each other. SpO2 reflects oxygenation, while tcPCO2 reflects ventilation; the first can still be normal while the second may herald early changes in respiratory status. Capnography may provide the earliest indication of opioid-induced respiratory depression. It is important to monitor changes from a baseline tcPCO2 level. As the tcPCO2 level starts to increase, early intervention and changes in medication can be made.

The present study aims to examine combined oxymetry and transcutaneous capnography using a single earlobe sensor (V-Sign™, Sentec AG, Therwil, Switzerland) in chronic pain patients treated with opioids where non-invasive monitoring of ventilation is needed because ventilatory disturbances are suspected. This may, potentially, improve patient's quality of life.

DETAILED DESCRIPTION:
1. Aim of study 1.1 Background

   Opioids are an effective instrument for patients with acute and chronic pain. Their route of administration ranges from transdermal to subcutaneous application through to Intravenous Patient-Controlled Analgesia (IV-PCA).

   The use of IV-PCA-pumps has considerable advantages including decreased delay in the administration of opioids from the time requested, individual dose intervals, self -control of their therapy, rapidity and ease of dose titration . These potential benefits, however are balanced by the need for careful assessment of adverse effects, including decreased quality of life because of the patient's sedation, constipation and possible episodes of bradypnoea and desaturation, eventually leading to respiratory depression (RD) requiring treatment. Often described safety features that help prevent overdosing are PCA bolus dose, delay, and lockout interval.

   Even though the risk of serious, potentially life threatening complications by using IV-PCA without a background infusion was described to be very low (0.24%) compared to other methods of opioid delivery , adverse effects like worrying degrees of hypoxemia and bradypnoea do occur and often remain undetected due to the lack of continuous monitoring. One of the possible causes of patient harm are medication errors associated with PCA administration, a common form of PCA errors, which is a significant source of preventable patient morbidity and hospital resource utilization.

   But not only patients with IV-PCA-pumps are at risk of harm, but all patients treated with opioids (distinguished by their formulations; oral, dermal, intravenous, short-acting, continuous-release) are due to the feared adverse effect of respiratory depression.

   It can be caused by a self-potentiating "vicious cycle" which may result in respiratory arrest: Hypoventilation impairs gas exchange, resulting in increased carbon dioxide, decreased oxygen and pH (respiratory acidosis). In turn, suppression of the chemoreceptor responses to increased carbon dioxide levels reduces the normally protective central response which would increase breathing efforts.

   The individual patient response to a particular dose of opioids depends on diagnosed or unrecognized comorbidities. Clinical experience has shown that it is not possible to prospectively identify all patients who may be at increased risk.

   Conventional opioid monitoring protocol may fail to detect frequent episodes of bradypnoea and desaturation measured by the respiratory rate (RR) and Saturation of Peripheral Oxygen (SpO2) because even at a low respiratory rate SpO2 is usually maintained, so that pulse oxymetry might fail to detect respiratory deterioration, particularly if a patient is receiving supplemental oxygen.

   Therefore, continuous monitoring could be considered more sensitive, especially if it contains the measurement of Partial Pressure of Carbon dioxide (PCO2), which is a good parameter for monitoring ventilatory function. As the American Society of Anesthesiologists emphasizes, ventilation and oxygenation must be considered as separate physiologic processes. Ventilatory function is monitored by PCO2 whereas oxygenation is expressed through SpO2.

   Thus, even continuous monitoring of heart rate and SpO2 by pulse oxymetry is not a substitute for monitoring respiratory rate (RR) and PCO2. By capnographic monitoring patient's desaturation might be anticipated if a decrease in RR and thus rise of PCO2 level from baseline occurs. Hence, adjustment of medication doses can be made earlier and serious adverse events may be prevented.

   The 'gold standard' method to measure the arterial partial pressure of carbon dioxide (PaCO2) is still the arterial blood gas analysis. But arterial sampling including catheterization or intermittent arterial puncture is invasive and expensive and associated with pain and discomfort for the patient. Therefore cutaneous carbon dioxide tension (PcCO2) measurement was suggested to be used as a non-invasive surrogate measure of PaCO2.

   Transcutaneous measurement of CO2 (tcPCO2) is based on the observation that this gas has a high tissue solubility and diffusion through the skin. This permits the non-invasive measurement of the arterial PCO2. But despite increasing interest, the role of PCO2 as the real measure of respiratory function appears to be widely underestimated. The reason for PCO2 playing only a minor role may be referred to different causes: For many years measurement of tcPCO2 was inaccurate and impracticable with sensors being fragile and expensive, requiring frequent calibration and changing of skin site of the sensor to avoid thermal injury to the skin. But modern devices have features like automatic calibration, shorter response and equilibration times.

   Combined cutaneous capnography (tcPCO2) and oxymetry (SpO2) can now be gathered by a single earlobe sensor. Based on the Severinghaus principle , tcPCO2 is measured by a sensor with a heated surface electrode on the skin. The local hyperaemia induces an increase of arterial blood in the dermal capillary bed under the sensor. The usefulness of this method is limited in some clinical situations including profound peripheral vasoconstriction or circulatory centralization in shock or skin edema. Chhajed et al. could show a good agreement between values obtained by using combined oxymetry and transcutaneous capnography with arterial blood gas analyses in a large study sample.

   In conclusion, SpO2, and tcPCO2, are important clinical parameters that should be used in conjunction with each other. SpO2 reflects oxygenation, while tcPCO2 reflects ventilation; the first can still be normal while the second may herald early changes in respiratory status. Capnography may provide the earliest indication of opioid-induced respiratory depression. It is important to monitor changes from a baseline tcPCO2 level. As the tcPCO2 level starts to increase, early intervention and changes in medication can be made.

   The present study aims to examine combined oxymetry and transcutaneous capnography using a single earlobe sensor (V-Sign™, Sentec AG, Therwil, Switzerland) in chronic pain patients treated with opioids where non-invasive monitoring of ventilation is needed because ventilatory disturbances are suspected. The Sentec Monitoring System is already in use for years in clinical settings, for instance: Neonatology, Pneumology and Surgery, etc.

   The intention of this study is to prove the feasibility for using this sensor in a hospital setting which may allow avoiding oversedation leading to decreased activity and other troublesome adverse effects. This may, potentially, improve patient's quality of life.

   1.2 Specific aims

   We want to show that continuous monitoring using combined transcutaneous capnography and oxymetry allows for a better support for patients treated with opioids for chronic pain regarding pain quality and possible adverse events. Furthermore we want to use this study as a feasibility trial to generate new hypotheses for possible future studies.

   1.3 Hypothesis

   Continuous monitoring of tcPCO2 and SPO2 may help to warrant for a better support of patients with opioid administration by a minimal additional effort. In the end an effective monitoring shall contribute to enhance therapy control and therefore increase both patient's safety and quality of life.
2. Study design

This study will be used as a Feasibility Trial for possible future studies. Our primary objective is to investigate whether continuous monitoring by using the SenTec Monitoring System is feasible in patients with opioid administration.

2.1 Study Procedures

We plan to consecutively recruit patients who need for their pain control the IV-PCA, transdermal, oral or subcutaneous opioids and are hospitalized in the Hildegard Hospital in Basel, Switzerland. Recruitment of patients will start June 2012 and will end as soon as 30 patients are recruited (at the latest in September 2013)

30 patients needing IV-PCA, subcutaneous, transdermal or oral Opioids for their pain control, will be conventionally monitored during 24 hours after having filled out the informed consent form. Care workers will record principal and secondary diagnosis, measure respiratory rate (RR), note quantity and name of consumed opioids, record serious adverse events requesting antagonists, cardiopulmonary resuscitation (CPR) or death and inquire for common adverse effects in opioid therapy such as sedation, pruritus, nausea/vomiting, dryness of the mouth, dizziness, myoclonus, constipation, fatigue, sweating, confusion and hallucinations. All patients will qualify their pain using the McGill Pain Questionnaire (MPQ) as well as quantify their pain with the aid of a Numeric Rating Scale (NRS).

For the subsequent 48h all patients will continuously be monitored by a single earlobe sensor (SenTec Monitoring System) in addition to the measurements/ questionnaires described above. Furthermore nurse's ratings of the additional time expense caused by the use of the SenTec Monitoring System will be recorded using a NRS.

3 Selection and Withdrawal of Subjects 3.2 Recruitment of patients

Patients treated with an IV-PCA and other application forms of opioids such as transdermal or subcutaneous opioid-administration for chronic pain who are hospitalized in the Hospital Hildegard, Basel, Switzerland, will be approached by a member of our study team. Patients are not only terminal Patients but as well Patients that are hospitalized for adjustment of pain medication and are going to be discharged. Participation in this study is voluntarily and the participating subjects will not be advantaged.

3.1 Subject Inclusion Criteria

* Older than 18 years
* Capable of giving informed consent
* Needing opioids (oral, transdermal, subcutaneous, IV-PCA) for pain control (opioid naïve or patients on chronic opioid therapy ) 3.2 Subject exclusion criteria
* No consent for participation
* Absence of power of judgment 3.3 Subject Withdrawal

In case a subject decides to discontinue our study for personal reasons, the withdrawal will be documented on the CRF (case report form) of the patient and another patient will be recruited to replace the study drop-out.

4 Measures and Questionnaires

4.1 SenTec Digital Monitoring System

The SenTec Digital Monitoring System allows a continuous and non-invasive monitoring of carbon dioxide tension (PCO2), functional oxygen saturation (SpO2) and pulse rate. The portable patient monitor receives its signals over a cable adapted to a specific sensor (V-Sign™ Sensor) and sends it to a remote monitoring station and secondary alarm surveillance (V-CareNeT™). The signal will be forwarded additionally to a mobile application which is at the time designed and developed.

The combined digital SaO2/PcCO2 sensor unifies the elements of an electrochemical Severinghaus-type carbon dioxide tension sensor with a conventional, reflectance 2-wave-length pulse oxymetry which allows a noninvasive and continuous estimation of arterial carbon dioxide tension and oxygen saturation.

This method to measure CO2 potentiometrically by determining the pH of electrolyte layer separated from the skin by a highly permeable membrane was described by Severinghaus and Bradley. The sensor is warmed to a constant surface temperature of 42.0°C to improve local arterialization and, hence, diminish the arterio-venous PCO2 difference and increase gas diffusion. Regular recalibration is mandatory for optimal transcutaneous signals and is known as a limiting factor. At this occasion skin surface will be inspected to avoid local side-effects. Sensors can be safely kept continuously for periods of up to 8 h with minimal risk of thermal skin injury. In case of further continuance in position the sensor will be programmed to trigger an alarm message and to cool down to 39.0°C automatically after 15 minutes (a total of 8h 15 min) if the alarm hasn't been switched off in time.

For subsequent analysis measurements will consecutively be downloaded from the SenTec Digital Monitoring System using V-STATS™ PC Software. The maximum period of measuring will be 3 days.

4.2 Numeric Rating Scale (NRS)

The use of pain scales as the Numerical Rating Scale (NRS) is recommended for assessment of pain intensity based on self- report. The NRS is an 11-point scale consisting of integers from 0 (no pain) through 10 (pain as bad as you can imagine). Respondents then select the single number that best represents their pain intensity. An advantage of NRS is that incorrect responding does not appear to be associated with persons at risk for cognitive difficulties such as some elderly individuals or persons on high doses of opioid analgesics.

Furthermore nurses ratings of the additional time expense by using the SenTec Monitoring System will be gathered by using the NRS (0 = no additional effort, 10 = maximal additional effort).

4.3 Adverse effects

Common adverse effects of opioid therapy will be reported by asking the patients themselves if they feel bothered by pruritus, nausea, dryness of the mouth, dizziness, myoclonus, constipation, fatigue, sweating, confusion and hallucinations (answer yes/no). Depth of sedation will be recorded by the nurses.

4.4 McGill Pain Questionnaire (MPQ)

The McGill Pain Questionnaire was designed in 1975 for the use in pain patients to specify sensory, affective and evaluative dimensions of subjective pain experience. It provides quantitative information that can be treated statistically and is supposed to be sufficiently sensitive to detect differences among different methods to relieve pain. In 1988 a German version of the McGill Pain Questionnaire has been developed.

4.5 Respiratory Depression

Assessment of respiratory status goes hand in hand with sedation assessment. The nurse should watch the rise and fall of the patient's chest to determine the rate, depth, and regularity of respirations. There is no consensus on definition of a clinically significant respiratory depression. Clinical significance is featured by a decrease in rate and depth from patient's baseline respiratory status. We define respiratory depression as a decrease of respiratory rate on less than 8 breath per minute and/or PtcCO2 ≥ 6.0 kPa (≥45mmHg).

4.6 Serious adverse events and complications

Serious adverse events necessitating intervention such as the use of antagonists, positive pressure ventilation, cardiopulmonary resuscitation (CPR) or death will be noted.

4.7 Quantity of consumed opioids

The quantity of consumed opioids during measuring time will be recorded noted in [mg]

4.8 Advantage and disadvantage for nursing staff

Nursing staff will be asked to declare gain and further efforts caused by additional monitoring using Sentec Monitoring System.

5 Statistical Plan

5.1 Primary and Study Endpoints

Primary Endpoint

- Number of events of respiratory depression (PtcCO2 ≥ 6.0 kPa (≥45mmHg) and/or a decrease of respiratory rate on less than 8 breaths per minute) after 48 h of measuring by Sentec Monitoring System

Secondary Endpoints

* Quantity and quality of pain
* Incidence of adverse effects (sedation, pruritus, nausea, dryness of the mouth, dizziness, myoclonus, constipation, fatigue, sweating, confusion and hallucinations)
* Serious adverse events and complications (use of antagonists, positive pressure ventilation, cardiopulmonary resuscitation (CPR), death)
* Amount of delivered/ demanded doses of consumed opioids
* Nurses' additional time expense by using the SenTec Monitoring System
* Nurses' contentment with the additional Monitoring using SenTec Monitoring System 5.2 Sample size and justification

We intend to include 30 individuals 5.3 Data analysis

* Primary and secondary diagnosis
* Stored data will be analyzed by specifically designed computer software (V-STATS™ PC Software)
* Numeric Rating Scale: Value (min =0, max = 10)
* Adverse effects: Number of each different effect (cumulated percentage of each one)
* McGill: 3 data sets (Numbers of words chosen, Pain rating index-(score), pain rating index-(rating)
* Respiratory Depression: Number and severity of events
* Severe adverse events and complications: Number and severity of each different event (cumulated percentage of each one)
* Quantity of consumed opioids: Total amount in [mg] (morphine equivalents) 5.4 Statistical analysis

Statistical significance will be acquired if a p value of less than 0.05 is attained.

5.5 Handling of missing values/censoring/discontinuations

Missing data will be minimized as far as possible by careful trial planning and conducting.

6 Study Management and Administration

6.1 Adherence to Protocol

The study will be conducted in compliance with the approved protocol. In case of any significant deviations from the study protocol the investigator will send an amendment for further approval to the Ethical Committee EKBB.

6.2 Data Collection and Protection

To collect "bed side" data a computer generated paper sheet containing the name and date of birth of the subject will be used. This data will be transferred to a CRF (case report form) and in doing so rendered anonymous before statistical analysis will be performed. Subsequently data transfer will be controlled by at least one person.

6.3 Archiving and Data Retention

All study-related records, such as CRFs, medical records, informed consent documents, information regarding participants who discontinued, and other pertinent data will be maintained and therefore retained as long as required by the applicable Swiss regulatory requirements (10 Years).

6.4 Direct Access to Original Data

The investigator (s) will provide the study related monitoring visits, audits and regulatory inspections for direct access to all data acquired.

6.5 Finances and Insurance

The Investigator declares that he has taken out an insurance policy for the total study length, covering the participants in respect of the risks involved in this study.

Study participants will receive no financial compensation for participation in this study.

7 Ethical Consideration 7.1 Subjects Information and Consent

All participating subjects will receive a consent form describing the study to help the subjects to make an informed consent about their participation in this study. Only after signing the consent form the subject will be submitted to any study procedure.

This consent form that will be used is submitted with this protocol for approval by the EKBB.

7.2 Risks and benefits for study participants

Patients aren't exposed to any risk by participating in this study. In case of upward trend of the tcPCO2 detected by the SenTec Monitoring System or a decrease of the patient's respiratory rate leading to a possible future respiratory depression, dosage of opioids may be adjusted according to the responsible physician's prescription.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Capable of giving informed consent
* Needing opioids (oral, transdermal, subcutaneous, IV-PCA) for pain control (opioid naïve or patients on chronic opioid therapy )

Exclusion Criteria:

* No consent for participation
* Absence of power of judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pain patients treated with opioids
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of events of respiratory depression and/or respiratory Depression | 48 h
  -Number of events of respiratory depression (PtcCO2 ≥ 6.0 kPa (≥45mmHg) and/or a decrease of respiratory rate on less than 8 breaths per minute) after 48 h of measuring by Sentec Monitoring System

SECONDARY OUTCOMES:
Quantity and quality of pain | 48 h
  quality of pain measured using VAS
Work quality For Nursing staff | 48 h
  * Nurses' additional time expense by using the SenTec Monitoring System
  * Nurses' contentment with the additional Monitoring using SenTec Monitoring System
Amount of delivered/demanded doses of consumed opioids | 48 h
Incidence of adverse effects | 48h
  sedation, pruritus, nausea, dryness of the mouth, dizziness, myoclonus, constipation, fatigue, sweating, confusion and hallucinations

CONTACTS AND LOCATIONS:
Locations (1):
- University clinic of internal medicine, Cantonal Hospital Baselland, Liestal, Basel-Landschaft, Switzerland